CLINICAL TRIAL: NCT04883554
Title: Impact of an Olfactory Sensory Therapeutic Group in the Therapeutic Armamentarium for Adolescent Patients With Restrictive Anorexia Nervosa, Pilot Study
Brief Title: Impact of an Olfactory Sensory Therapeutic Group for Adolescent Patients With Restrictive Anorexia Nervosa , Pilot Study
Acronym: Sens'Orality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-HPNCL-02
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Mind-Body Therapies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olfactory therapy group (Experimental): The therapeutic group takes place in specific stages on a weekly basis and lasts approximately 45 minutes. The group consists of a maximum of 6 patients of approximately the same age. The therapists leading the therapeutic group choose in advance the smells that will be offered to patients, based on one odor for each of the following categories: food and woody / flowery. The odors circulate between the participants of the group (patients and therapists), on wipes of blotting paper soaked in the bottles and soaked in the odors. The first step of the therapeutic group is "olfactory perception": this is the moment when the odors selected for the session are presented to the patients. Each scent goes around the patients and therapists, three times and without verbalization. Therefore, patients can express their feelings through drawing or writing on distributed sheets. .
  In a second step, called "rendering", patients are asked to express what they think of the smell presented.
  Interventions: Other: Olfactory therapeutic
- Body therapy group (Active Comparator): The therapeutic group takes place according to very specific stages at a weekly frequency and lasts 1 hour. The group is made up of a maximum of 6 patients.
  This workshop includes three times divided equally over a period of 1 hour:
  Kinesic time or time to set the body in motion (20 min):
  These techniques involve lying on the floor on a mat and approaching the movement slowly. The movements are suggested by the patients and then imitated by the rest of the group.
  Kinesthetic time: time of slow movements (20 min):
  During this time, the patient is asked to find a period of calm close to immobility without imposing the instruction. They are asked to touch the different parts of the body as slowly as possible in isolation, starting and ending in the center of the body.
  Talk time (20 min):
  Patients are invited to verbalize what they felt bodily
  Interventions: Other: Body therapy

INTERVENTIONS:
Other: Olfactory therapeutic — The sessions of the olfactory sensory therapy group take place according to the care framework at a frequency of one session of 45 minutes per week
  Arms: Olfactory therapy group
Other: Body therapy — very specific stages at a weekly frequency and lasts 1 hour. Kinesic time or time to set the body in motion (20 min) Kinesthetic time: time of slow movements (20 min) Talk time (20 min)
  Arms: Body therapy group

SUMMARY:
Anorexia nervosa is a severe eating disorder of multifactorial origin and for which there is, to date, no specific, standardized and protocolized management for anorexic patients or data on the superiority of anorexia. type of psychotherapy. The literature reports altered olfactory capacities in anorexia nervosa and the effectiveness of sensory-mediated therapies in several mental disorders.

This prospective, single-center, randomized and controlled study proposes the evaluation of the therapeutic impact of an olfactory sensory group carried out during the specialized care of patients aged 12 to 20 years, with anorexia. The main objective is to compare the clinical course of eating disorder, using the Eating Attitudes Test-40 (EAT-40) scale score performed at study inclusion and at 9 months at 9 months, of patients participating in an olfactory sensory therapeutic group compared to a body approach therapeutic group.

The secondary objectives of this study are to compare between a treatment associated with an olfactory sensory therapeutic group and a body approach therapeutic group, the evolution of the Body Mass Index at 9 months, overall functioning, evolution of cognitive and sensory capacities, and evolution of the therapeutic alliance at 9 months

DETAILED DESCRIPTION:
Currently, there is no specific consensus on the treatment of anorexia nervosa due to a lack of international scientific evidence. The guidelines recommend that patients be managed on an outpatient basis whenever possible with psychological treatment. This treatment must be provided by experience and a qualified service that can also assess the physical risks. Family therapy is the most popular psychological treatment for children and adolescents with anorexia nervosa. The drugs are considered adjunctive therapy and often have not shown significant results. Nutritional rehabilitation programs establish target weights based on body mass index (BMI). The target is calculated for the age percentiles. Weight restoration requires cognitive restructuring therapy to treat cognitive impairment associated with a state of calorie restriction. In the University Department of Child and Adolescent Psychiatry (UDCAP), we offer highly specialized treatment for restrictive anorexia in children and adolescents, which has been progressively developed over more than 25 years by a multidisciplinary team based on sensory-cognitive therapy is associated with this specific treatment. This treatment, based on sensori-cognitive therapy, is combined with the specific treatment recommended by theFrench National Authority for Health (HAS :Haute Autorité de Santé). The literature hypothesizes impaired sensory abilities are a central symptom of anorexia nervosa. Therefore, sensory impairment is expected to alter instinctive perceptions and gradually destroy recognition of primary needs. This theory of sensory integration is based on the principles of neuroscience, psychology and rehabilitation. Stimulation of olfactory sensory cognition has been used systematically in the first-line treatment of anorexic patients at UDCAP for many years and has shown encouraging clinical results which remain to be scientifically demonstrated. This study proposes the evaluation of the therapeutic impact of an olfactory sensory group carried out during the specialized care of patients with anorexia.

The main objective of this single-center, randomized, controlled, single-blind, prospective study is to compare the clinical course of eating disorder at 9 months of patients participating in an olfactory sensory therapeutic group compared to a body approach therapeutic group, classically recommended in conventional management, in patients aged 12 to 20 years with restrictive anorexia nervosa. The main objective is assessed using the Eating Attitudes Test-40 (EAT-40) scale score performed at study inclusion and at 9 months. The secondary objectives of this study are to compare between a treatment associated with an olfactory sensory therapeutic group and a body approach therapeutic group : The evolution of the Body Mass Index (BMI) at 9 months, Overall functioning, assessed using the Clinical Global Impression (CGI) at 9 months, Clinical evolution at 9 months assessed with clinical scales : Quality of life deterioration score (QUAVIAM), Beck Depression Inventory (BDI), Situational anxiety and anxiety trait inventory (STAI-Y), Yale-Brown Obsession Compulsion Scale (Y-BOCS), Child Post-Traumatic Stress-Reaction Index (CPTS-RI), The Autistic Quotient (AQ) ; Evolution of cognitive and sensory capacities at 9 months assessed with mental flexibility tests of Cognitive Remediation Therapy (CRT) and the self-questionnaire "Sensory profile" (Brown, Dunn)., Evolution of the therapeutic alliance at 9 months will be assessed with the Helping Alliance Questionnaire (HAQ).

The number of subjects required is 30 patients, 15 patients per group, with alpha risk of 5% and a power of 80%, with an estimated number of lost to follow-up of 30%.

The estimated duration of this study is 27 months, with a participation time for each patient of 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 12 to 20 years old
* Diagnosed with restrictive anorexia nervosa, according to Diagnostic and Statistical Manual 5 (DSM 5) criteria and who have not yet entered the care pathway
* Affiliated with the social security scheme
* Good understanding of written and oral French
* Collection of informed consent from the adult subject
* Collection of informed consent from one of the two parents or holder of parental authority if the subject is a minor

Exclusion Criteria:

* All pathologies that may explain an olfactory sensory disorder: genetic, neurological, neurosensory or rhino laryngeal pathologies (chronic bronchitis, polyps, etc.)
* History of participation in an olfactory sensory therapy group
* The restriction disorder or avoidance of food intake (ARFID, Avoidant and Restrictive Food Intake Disorder)
* Active smoking
* Intellectual disability (ITQ <70)
* Known allergy to essential or fragrant oils
* A urine pregnancy test will be performed for young women of childbearing age.
* Persons deprived of their liberty by a judicial or administrative decision, persons undergoing psychiatric treatment by virtue of ..
* Adults who are the subject of a legal protection measure or who are unable to express their consent.
* Foreseeable inability to comply with the instructions defined and exposed upon inclusion

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
evolution of eating disorder | at 9 months after inclusion
  Clinical course of the eating disorder of anorexic patients scores of the Eating Attitudes Test-40 (EAT-40) scale.
  Self-diagnostic and quantitative questionnaire of 40 questions 6 response levels ranging from: not at all / never to extremely / always Items 1, 18, 19, 23, 27, 34, 39 are presented inverted. Whatever the direction of the presentation, each extreme response of the anorexic type corresponds to 3 points, the next to 2, the third to 1 and the three others to 0.
  The score varies from 0 to 120. The threshold score is 30, that is, any subject with a score ≥ 30 has an eating disorder Performed at inclusion of subjects in the study and at 9 months

SECONDARY OUTCOMES:
Evolution of the Body Mass Index (BMI) | at 3, 6, and 9 months after inclusion
  Weightings carried out in the morning, on an empty stomach on the undressed subject.
  - BMI performed at the inclusion and at 3, 6, and 9 months
Clinical Global Impression (CGI) Severity scale | at 9 months after inclusion
  Allow a clinician to assess the improvement in a patient's condition over time, after prescription of treatment or after discontinuation, to assess overall functioning at 9 months.
  Number of items for questionnaire: 7
  the "CGI Severity Scale", the examiner rates the severity of the patient's clinical condition using a seven-point scale.
  Performed at the inclusion and at 9 months. A continuous analysis of the results of this scale will be retained. An decrease in scores measured before and after the therapy group means an improvement
Clinical Global Impression (CGI) Improvement scale | at 9 months after inclusion
  Allow a clinician to assess the improvement in a patient's condition over time, after prescription of treatment or after discontinuation, to assess overall functioning at 9 months.
  Number of items questionnaire: 7
  During follow-up, with the "CGI Improvement Scale", the doctor assesses on a seven-point scale the improvement in the patient's clinical condition following treatment.
  Performed at the inclusion and at 9 months. A continuous analysis of the results of this scale will be retained. An decrease in scores measured before and after the therapy group means an improvement
Quality of life deterioration score (QUAVIAM) | at 9 months after inclusion
  Evaluates the quality of somatic, psychological, socio-professional, hedonic and related to eating disorder.
  Number of items: 61 Score from 0 to 610 Each item can be rated from 0 to 10. A decrease in scores measured before and after the therapy group means an improvement
Beck Depression Inventory (BDI) | at 9 months after inclusion
  Self-diagnostic questionnaire allowing a quantitative estimate of the intensity of depressive symptoms.
  Number of items: 21 scored from 0 to3 Total score from 0 (no depressive symptoms) to 63 (severe depression) A continuous analysis of the results of this scale will be retained. An increase in scores measured before and after the therapy group means an improvement.
Situational anxiety and anxiety trait inventory (STAI-Y) | at 9 months after inclusion
  This self-diagnostic questionnaire aims to assess anxiety as a personality trait and anxiety as an emotional state related to a particular situation.
  Number of items: 20 items for each questionnaire The rating scale varies from 1 (almost never) to 4 (almost always). A continuous analysis of the results of this scale will be retained. A decrease in scores measured before and after the therapy group means an improvement
Yale-Brown Obsession Compulsion Scale (Y-BOCS) | at 9 months after inclusion
  In the form of a structured interview that provides a measure of the severity of obsessive symptoms.
  The interview is divided into three successive stages:
  1. Define obsessions and compulsions, then use the past and current obsessions and rituals checklist.
  2. Define the three main haunting thoughts, the three main motor rituals, the three main situations avoided.
  3. Rate the dimensions for obsessions and compulsions from 0 to 4. Number of items: 10 It makes it possible to distinguish an obsession score (from 0 to 20) and a compulsion score (from 0 to 20).
  Depending on the total score obtained, we will distinguish:
  * A score of 0 to 7 is considered non-clinical
  * A score of 8 to 15 is considered light
  * A score of 16 to 23 is considered moderate
  * A score of 24 to 40 is considered severe. A continuous analysis of the results of this scale will be retained. A decrease in scores measured before and after the therapy group means an improvement.
Child Post-Traumatic Stress-Reaction Index (CPTS-RI) | at 9 months after inclusion
  Self-administered questionnaire used to assess the severity of post-traumatic reactions.
  He begins with a general question asking if he has ever experienced an event that he found traumatic.
  Number of items: 20 The child responds to each item on a 5-point Likert scale, ranging from 0 (never) to 4 (most of the time). The scores for the 20 items are added together, for a total score between 0 and 80.
  The following cut-off points can be used to determine the severity of post-traumatic stress reactions: 0-11 (unlikely), 12-24 (mild), 25-39 (moderate), 40-59 (severe), and 60-80 (profoundly serious) (73).
  A decrease in scores measured before and after the therapy group means an improvement.
The Autistic Quotient (AQ) | at 9 months after inclusion
  This self-administered questionnaire aims to assess autistic traits in people of average or better intelligence.
  Number of items: 50 The responses "strongly agree" and "somewhat agree" are scored 0 and the responses "somewhat disagree" and "not agree at all" are graded 1. The maximum total score is 50 and autistic functioning is retained from the threshold score of 30.
  A decrease in scores measured before and after the therapy group means an improvement
Cognitive Remediation Therapy (CRT) | at 9 months after inclusion
  mental flexibility tests measure the evolution of cognitive abilities; performed at the inclusion and at 9 months.
  the measure is done with three tasks :
  * The Stroop: assesses subjects alternating between different aspects of the same stimulus or between different instructions for the same task, quickly and correctly
  * test of Tangled words: The purpose is to locate, in a grid filled with letters, words known in the dictionary, read in both directions, horizontally, vertically and diagonally.
  * test of entangled words: The goal is to identify the words of a proposed topic among irrelevant words.
  The time required for the subject to complete the tasks will be measured within a time limit of no more than 8 minutes.
  A reduction in the processing time after participating in the therapeutic workshops means an improvement.
  A continuous analysis of the results of this scale will be retained.
"Sensory Profile" self-quiz (Brown, Dunn). | at 9 months after inclusion
  This self-administered questionnaire aims to measure the evolution of sensory abilities.
  Number of items: 60
  Response scores range from 1 for "almost never" to 5 for "almost always". This questionnaire assesses the subject's sensory cognitive abilities according to categories whose scores vary between 15 and 75:
  * Weak recording: items 3, 6, 12, 15, 21, 23, 36, 37, 39, 41, 44, 45, 52, 55, 59
  * Sensory research: items 2, 4, 8, 10, 14, 17, 19, 28, 30, 32, 40, 42, 47, 50, 58
  * Sensory sensitivity: items 7, 9, 13, 16, 20, 22, 25, 27, 31, 33, 34, 48, 51, 54, 60
  * Avoidance of sensations: items 1, 5, 11, 18, 24, 26, 29, 35, 38, 43, 46, 49, 53, 56, 57
  A continuous analysis of the results of this scale will be retained. Performed at the inclusion and at 9 months.
Helping Alliance Questionnaire (HAQ) | at 9 months after inclusion
  This self-administered questionnaire aims to evaluate the therapeutic alliance. Number of items: 13 Each item is rated on a 6-point Likert scale ranging from 1 "Strongly Disagree" to 6 "Strongly Agree". Scores range from 13 to 78.
  Performed at the inclusion and at 9 months. A continuous analysis of the results of this scale will be retained. An increase in scores measured before and after the therapy group means an improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice, France